CLINICAL TRIAL: NCT02712606
Title: A Study About Accuracy of Pulse Oximeter With Hypoxemic Measurements (Blue Sensor) in Children With Cyanotic Congenital Heart Disease
Brief Title: Accuracy of Pulse Oximeter With Hypoxemic Measurements
Acronym: bluesensor
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, professor, Seoul National University Hospital
Other Study IDs: H-1602-060-740
Record Dates: First submitted 2016-03-09; First posted 2016-03-18 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Cyanotic Congenital Heart Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
A study about accuracy of pulse oximeter with hypoxemic measurements (Blue sensor, Masimo, Irvine, CA, USA) in children with cyanotic congenital heart disease

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of cyanotic congenital heart disease
* weight 2.5kg to 30kg
* undergoing general anesthesia
* preoperative SpO2<97%

Exclusion Criteria:

* none

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: tertiary care university children's hospital
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2016-03; Primary Completion 2017-03 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
accuracy of pulse oximetry using blue sensor | From the start of anesthetic induction until discharge from hospital, assessed up to 1 week.
  Each arterial blood gas sample and pulse oximeter oxygen saturation (SpO2) from blue sensor pulse oximetry are simultaneously obtained if the SpO2 is <97%.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea